CLINICAL TRIAL: NCT06101134
Title: A Phase 2 Open-label, Two-cohort Study to Evaluate Patient Preference for Nivolumab + Relatlimab Fixed-dose Combination Subcutaneous Versus Nivolumab + Relatlimab Fixed-dose Combination Intravenous and Nivolumab Subcutaneous Versus Nivolumab Intravenous in Participants With Melanoma
Brief Title: A Study to Evaluate Whether Participants With Melanoma Prefer Subcutaneous vs Intravenous Administration of Nivolumab and Nivolumab + Relatlimab Fixed-dose Combinations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-1044; U1111-1289-5947 (Other: WHO); 2023-504515-33-00 (Other: EU CTR)
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Melanoma
Keywords: Patient preference; Nivolumab Relatlimab IV; Nivolumab Relatimab SC; Melanoma; rHuPH20; FDC IV; FDC SC; Adjuvant; Metastatic; Switch; Nivolumab; Relatlimab
MeSH Terms: conditions — Melanoma; Patient Preference; Neoplasm Metastasis | interventions — Opdualag; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Metastatic Melanoma (Experimental)
  Interventions: Drug: relatlimab+nivolumab; Drug: relatlimab+nivolumab+rHuPH20
- Cohort 2: Resected Melanoma (Experimental)
  Interventions: Drug: nivolumab; Drug: nivolumab+rHuPH20

INTERVENTIONS:
Drug: relatlimab+nivolumab — Specified dose on specified days
  Other Names: BMS-986213; Opdualag
  Arms: Cohort 1: Metastatic Melanoma
Drug: relatlimab+nivolumab+rHuPH20 — Specified dose on specified days
  Arms: Cohort 1: Metastatic Melanoma
Drug: nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Cohort 2: Resected Melanoma
Drug: nivolumab+rHuPH20 — Specified dose on specified days
  Other Names: BMS-986298
  Arms: Cohort 2: Resected Melanoma

SUMMARY:
The purpose of this study is to assess the patient's preference for nivolumab subcutaneous (SC) or nivolumab + relatlimab fixed-dose combination (FDC) SC and provide patient experience data by route of administration. This study will also generate safety data which will further characterize the safety profile of patients switching the route of administration from intravenous (IV) to SC.

ELIGIBILITY:
Inclusion Criteria:

* Must have either metastatic melanoma and have not had previous treatment for their cancer, or resected melanoma and have had the cancer removed fully with surgery no later than 12 weeks before the start of treatment and confirmed free of disease
* Must have a low level of disability and cancer that is considered advanced for metastatic melanoma and at risk for becoming advanced (intermediate) or advanced for resected melanoma

Exclusion Criteria:

* Must not have any brain cancer/disease treated with radiation, any cancer in the eyes or mucous membranes (cells that cover inside surface of parts of the body and keep it moist), any autoimmune disease, or any condition that is being treated with steroids for inflammation (corticosteroids) or medication to decrease the body's immune system response (immunosuppressive drugs)

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants that prefer subcutaneous (SC) route of administration as assessed by Question 7 of the Patient Experience and Preference Questionnaire (PEPQ) | At Cycle 4 Day 1 (each cycle is 28 days)

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to approximately 2.5 years
Number of participants with Serious AEs (SAEs) | Up to approximately 2.5 years
Number of participants with treatment-related AEs | Up to approximately 2.5 years
Number of participants with AEs leading to discontinuation | Up to approximately 2.5 years
Number of participants with Immune-mediated AEs (IMAEs) | Up to approximately 2.5 years
Number of participants with other events of special interest (OESIs) | Up to approximately 2.5 years
Number of participants with injection/infusion-related AEs | Up to approximately 2.5 years
Number of deaths | Up to approximately 2.5 years
Number of participants with laboratory abnormalities | Up to approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (9):
  - Local Institution - 0007, Anchorage, Alaska
  - Local Institution - 0013, Phoenix, Arizona
  - Local Institution - 0010, San Francisco, California
  - Local Institution - 0034, Atlanta, Georgia
  - Local Institution - 0032, Edgewood, Kentucky
  - Local Institution - 0028, Albuquerque, New Mexico
  - Local Institution - 0037, Edmonds, Washington
  - Local Institution - 0036, Issaquah, Washington
  - Local Institution - 0030, Seattle, Washington
- Chile (2):
  - Local Institution - 0015, Las Condes, Santiago Metropolitan
  - Local Institution - 0005, Concepción
- Greece (6):
  - Local Institution - 0019, Thessaloniki, B
  - Local Institution - 0014, Athens, I
  - Local Institution - 0029, Marousi, I
  - Local Institution - 0023, Holargos, Athens
  - Local Institution - 0008, Piraeus
  - Local Institution - 0033, Thessaloniki
- Italy (7):
  - Local Institution - 0017, Bergamo, BG
  - Local Institution - 0035, Meldola, FC
  - Local Institution - 0018, Milan, MI
  - Local Institution - 0012, Padua, PD
  - Local Institution - 0021, Roma, RM
  - Local Institution - 0004, Torino, TO
  - Local Institution - 0026, Napoli
- Spain (7):
  - Local Institution - 0011, Barcelona, B
  - Local Institution - 0022, Barcelona, B
  - Local Institution - 0009, Cartagena, MU
  - Local Institution - 0020, Badalona
  - Local Institution - 0027, Cantabria
  - Local Institution - 0003, San Pedro Alcántara, Málaga
  - Local Institution - 0006, Seville

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06101134.html